CLINICAL TRIAL: NCT04754035
Title: A Multi-Center, Open Label, Uncontrolled, Phase 2a Clinical Trial Evaluating the Safety and Efficacy of the Addition of Ibrutinib to Venetoclax Through a MRD-guided Approach in Relapsed/Refractory Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Clinical Study With Ibrutinib and Venetoclax for Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia
Acronym: IMPROVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paolo Ghia (Other)
Responsible Party: Sponsor-Investigator, Paolo Ghia, Principal Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PS-CLL-002
Record Dates: First submitted 2017-07-07; First posted 2021-02-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Venetoclax will be administered, initially as single agent, orally once daily (QD), starting with 20 mg on Day 1, followed by weekly dose escalation up to 400 mg At Cycle 12 Day 1 Minimal residual disease (MRD) in the peripheral blood will be evaluated in patients with CR or PR by flow cytometry. All MRD negative subjects (defined as those with MRD level in the PB <10-4 in the PB and in the BM aspirate) will discontinue venetoclax at the end of Cycle 12. All MRD positive subjects (defined as those with MRD level in the PB >10-4) and patients with stable disease will continue venetoclax and start treatment with ibrutinib at the standard dose for CLL of 420 mg QD. Venetoclax will be administered until unacceptable toxicity or disease progression or for a maximum of 2 years and ibrutinib will be continued until unacceptable toxicity, confirmed MRD negativity, or disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- venetoclax + ibrutinib (Experimental)
  Interventions: Drug: Venetoclax; Drug: Imbruvica Oral Product

INTERVENTIONS:
Drug: Venetoclax — venetoclax 20 mg, 50 mg, 100 mg
Drug: Imbruvica Oral Product — Imbruvica 140 mg

SUMMARY:
This is a Phase 2a, multicenter, open-label uncontrolled study aimed at determining therapeutic benefits of the addition of ibrutinib to venetoclax in patients with relapsed/refractory CLL based on a MRD-guided approach.

DETAILED DESCRIPTION:
Venetoclax will be administered, initially as single agent, orally once daily (QD), starting with 20 mg on Day 1, followed by weekly dose escalation up to 400 mg, if well tolerated [Ramp-up Period, according to the modified Venetoclax schedule in Phase 2 and 3 clinical trials] and continued thereafter. At Cycle 12 Day 1, disease status, renal function and risk of bleeding will be assessed. Minimal residual disease (MRD) in the peripheral blood will be evaluated in patients with CR or PR by flow cytometry. All MRD negative subjects (defined as those with MRD level in the PB <10-4 in the PB and in the BM aspirate) will discontinue venetoclax at the end of Cycle 12 (i.e. Cycle 12 Day 28). All MRD positive subjects (defined as those with MRD level in the PB >10-4) and patients with stable disease without any contraindications to ibrutinib treatment will continue venetoclax and start treatment with ibrutinib at the standard dose for CLL of 420 mg QD. Venetoclax will be administered until unacceptable toxicity or disease progression or for a maximum of 2 years and ibrutinib will be continued until unacceptable toxicity, confirmed MRD negativity, or disease progression.

MRD will be assessed every 3 months starting 3 months after treatment initiation; MRD negativity at Cycle 12 Day 1 will be evaluated in PB BM aspirate.

Patients experiencing clinical disease progression will discontinue study treatment and will be followed up for survival status and subsequent anti-cancer therapy.

Inclusion criteria 1. Documented CLL requiring treatment according to the IWCLL criteria (Hallek et al. 2008) 2. Relapsed/refractory CLL patients who received at least 1 prior therapy 3. Adequate bone marrow function without transfusion < 2 weeks of screening as follows:

a. Absolute neutrophil count (ANC) ≥1.0 x 109/L (growth factors administration is allowed) b. Platelets ≥30 x 109/L. If thrombocytopenia due to BM involvement, platelets should be ≥ 20 x 109/L c. Hemoglobin value ≥8.0 g/dl exclusion criteria

1. Transformation of CLL to aggressive NHL (Richter's transformation or pro-lymphocytic leukemia)
2. Known central nervous system (CNS) involvement
3. Inadequate renal function: CrCl <30 mL/min
4. Previous treatment with BTK and/or BCL2 inhibitors (patients previously treated with PI3K inhibitors are eligible)
5. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
6. Requires the use of warfarin, marcumar, or phenprocoumon (potential drug-drug interaction increasing exposure of warfarin or phenprocoumon): low molecular weight drugs e.g. heparin are acceptable
7. Treatment, administration or consumption of any of the following within 3 days prior to the first dose of venetoclax (see also Appendix G).

   1. Strong Cytochrome P450 3A (CYP3A) inhibitors
   2. Moderate CYP3A inhibitors
   3. Moderate or strong CYP3A inducers
   4. PI3K inhibitors (e.g. Idelalisib);
   5. Grapefruit or grapefruit products
   6. Seville oranges (including marmalade containing Seville oranges)
   7. Star fruit
8. Known history of human immunodeficiency virus (HIV) or active with hepatitis B virus (HBV) or hepatitis C virus (HCV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
9. History of other malignancies, except:

   1. Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without current evidence of disease.

Updated International Workshop on CLL (IWCLL, Hallek et al. 2008) criteria will be used to determine rates of response and progression for patients with CLL with the modification to exclude lymphocytosis as an isolated criterion of progression in patients treated with agents inhibiting B-cell receptor signaling.

The primary endpoint objective response rate (MRD negativity) as well as secondary efficacy endpoints (e.g. ORR, PR, CR, PFS) will be derived from Investigator assessment.

Patients who reach a complete and partial response, as per standard criteria, will be investigated using MRD testing for molecular response categories as described in IWCLL.

The safety and tolerability of study drug treatments will be evaluated by means of AEs (incidence and severity), performance status, physical examinations, 12-lead resting electrocardiograms (ECGs), and laboratory safety evaluations.

Laboratory and AE toxicities will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.

biomarker assessment

* Whole exome sequencing on leukemic samples before, during and after treatment and/or at relapse in order to dissect mechanisms of resistance.
* High-throughput sequencing for MRD detection
* Biochemical assays on the circulating leukemic population during ibrutinib treatment to study activation of signaling pathways.

Statistical considerations According to optimal Simon Two-Stage Phase 2 design, with the null hypothesis (P0) of a MRD-negative CR at 12 months of 5%, this study will consider a satisfactory efficacy of the venetoclax + ibrutinib combination worth of further investigation a P1 corresponding to a MRD-negative CR of 30%. Considering a standard type I error (α) of 0.05 and a power of 95%, 29 MRD positive patients will be necessary for the expansion phase of the trial. A first step analysis will be implemented when 9 MRD positive patients have been enrolled and study will proceed to complete the planned accrual if at least 1/9 patients will obtain a MRD negative CR at 12 months after starting Ibrutinib. Considering that 5% of patients are expected to reach a MRD negative CR with venetoclax alone, the target population to be enrolled into the trial is 31 patients.

ELIGIBILITY:
Inclusion criteria

1. ≥ 18 years of age
2. Documented CLL requiring treatment according to the IWCLL criteria (Hallek M et al, 2008)
3. Relapsed/refractory CLL patients who received at least 1 prior therapy
4. Adequate bone marrow function without transfusion < 2 weeks of screening as follows:

   1. Absolute neutrophil count (ANC) ≥1.0 x 109/L (growth factors administration is allowed)
   2. Platelets ≥30 x 109/L. If thrombocytopenia due to BM involvement, platelets should be ≥ 20 x 109/L
   3. Hemoglobin value ≥8.0 g/dl
5. The patient has adequate renal and hepatic function per local reference laboratory reference ranges as follows:

   1. Renal: patient has a creatinine clearance (CrCl) ≥ 30 mL/min
   2. Hepatic: AST and ALT ≤ 3 × the upper normal limit (ULN) of institution's normal range and bilirubin ≤ 1.5 × ULN. Patients with AIHA and Gilbert's syndrome may have a bilirubin > 1.5 × ULN, but these conditions must be clearly documented in clinical records.
6. Female patients of childbearing potential and non-sterile male patients must practice at least one of method of birth control with partner(s) beginning with initial treatment administration and continuing to 30 days after the last dose of study treatment. Female of child bearing potential must have a negative serum pregnancy test upon study entry
7. Male patient must agree to refrain from sperm donation, from initial treatment administration until 90 days after the last dose of treatment
8. Ability to provide written informed consent and to understand and comply with the requirements of the study

Exclusion criteria

1. Transformation of CLL to aggressive NHL (Richter's transformation or pro-lymphocytic leukemia)
2. Known central nervous system (CNS) involvement
3. Inadequate renal function: CrCl <30 mL/min
4. Previous treatment with BTK and/or BCL2 inhibitors (patients previously treated with PI3K inhibitors are eligible)
5. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
6. Requires the use of warfarin, marcumar, or phenprocoumon (potential drug-drug interaction increasing exposure of warfarin or phenprocoumon): low molecular weight drugs e.g. heparin are acceptable
7. Treatment, administration or consumption of any of the following within 3 days prior to the first dose of venetoclax (see also Appendix G):

   1. Strong Cytochrome P450 3A (CYP3A) inhibitors
   2. Moderate CYP3A inhibitors
   3. Moderate or strong CYP3A inducers
   4. PI3K inhibitor (e.g. Idelalisib);
   5. Grapefruit or grapefruit products
   6. Seville oranges (including marmalade containing Seville oranges)
   7. Star fruit
8. Known history of human immunodeficiency virus (HIV) or active with hepatitis B virus (HBV) or hepatitis C virus (HCV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
9. Known hypersensitivity to one or more study drugs
10. Known bleeding disorders (e.g. von Willebrand's disease) or hemophilia
11. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
12. Major surgery within 4 weeks of the first dose of study drug
13. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach, or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
14. Any uncontrolled active systemic infection or infection requiring systemic treatment that was completed ≤7 days before planned treatment start date
15. Prior allogeneic stem cell transplant
16. Lactating or pregnant
17. Unable to understand the purpose and the risks of the study and to provide a signed and dated informed consent (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
18. History of other malignancies, except:

    1. Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without current evidence of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease | 4 years
  Minimal residual disease (MRD) negativity rate evaluated by multi-colour flow cytometry analysis (limit of detection 10-4) within the treatment period

SECONDARY OUTCOMES:
Complete response (CR) rate | 4 years
Progression-free survival (PFS) rate at 12 months | 1 year
Progression Free Survival (PFS) | 4 years
Overall response rate (ORR) | 4 years
Duration of response (DOR) | 4 years
Overall Survival (OS); | 4 years
Adverse events | 4 years
  Type, frequency, and severity of adverse events (AEs) and relationship of AEs
Proportion of premature withdrawals | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Ghia, Prof, Study Chair — San Raffaele Hospital
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

REFERENCES:
- [Derived] Scarfo L, Heltai S, Albi E, Scarano E, Schiattone L, Farina L, Moia R, Deodato M, Ferrario A, Motta M, Reda G, Sancetta R, Coscia M, Rivela P, Laurenti L, Varettoni M, Perotta E, Capasso A, Ranghetti P, Colia M, Ghia P. Minimal residual disease-driven treatment intensification with sequential addition of ibrutinib to venetoclax in R/R CLL. Blood. 2022 Dec 1;140(22):2348-2357. doi: 10.1182/blood.2022016901. PMID 35921541